CLINICAL TRIAL: NCT07007819
Title: Community-Engaged Behavioral Sleep and Circadian Intervention for School-Aged Children With Autism Spectrum Disorder
Brief Title: Community-Engaged Sleep Intervention for School-Aged Children With Autism Spectrum Disorder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: American Academy of Sleep Medicine (Other); National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Megan Wenzell, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY20240404
Record Dates: First submitted 2025-05-19; First posted 2025-06-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sleep Disturbance; Autism Spectrum Disorder
Keywords: Sleep and Circadian Intervention; Autism Spectrum Disorder; Pediatrics; Sleep Disturbance
MeSH Terms: conditions — Parasomnias; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The sleep and circadian intervention is guided by the Pediatric Sleep Health Framework that encourages improvement in six pediatric sleep dimensions (B-SATED): sleep behaviors; parents' satisfaction with child sleep; daytime alertness/sleepiness; appropriate timing of sleep within the 24-hour day; sleep efficiency, i.e., ease of falling and staying asleep; and sleep duration. The Sadeh and Anders Sleep-Wake Regulation Model was used to propose linkages between outcomes.
Who Masked: Outcomes Assessor
Masking Description: A trained researcher, masked to group assignment, will administer the primary outcome as an independent evaluator. Since this is a pilot study, the PI will deliver the intervention to allow for real-time adjustments and optimal quality control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Sleep and Circadian Intervention (Experimental): Up to 50 children will be randomly assigned (1:1) to the modified sleep and circadian intervention or enhanced usual care for 12 weeks.
  Interventions: Behavioral: Modified Sleep and Circadian Intervention
- Enhanced Usual Care Control Condition (Active Comparator): Up to 50 children will be randomly assigned (1:1) to the modified sleep and circadian intervention or enhanced usual care for 12 weeks.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Modified Sleep and Circadian Intervention — The modified sleep and circadian intervention has 5 individual sessions that will be delivered via Zoom to parents over 12 weeks and consists of 4 cross-cutting modules (functional analysis, goal setting, motivational interviewing, sleep education), 5 core sessions, and 7 optional modules that are delivered based on personalized treatment goals. The intervention format is as follows: (1) 60-minute session with consultation on setting goals and developing an action plan to improve sleep timing, quantity, and regularity; (2) 5-minute weekly follow-ups and a 3-night sleep diary; and (3) four 30-45-minute booster sessions every 3 weeks. Child attendance is optional.
  Arms: Modified Sleep and Circadian Intervention
Behavioral: Enhanced Usual Care — Enhanced Usual Care (EUC) is an active comparison treatment balanced for time and attention. Participants will be asked to maintain their typical sleep schedules. EUC sessions will review the interrelationships between stress, diet, health, exercise, and behavior, with a sleep education portion < 10 minutes and no encouragement to change behavior. EUC sessions will be used to establish rapport and promote study retention. EUC participants will not complete weekly sleep diaries. At the end of Week 12, EUC participants will receive a 1-hour optional Zoom session with the PI on sleep education.
  Arms: Enhanced Usual Care Control Condition

SUMMARY:
As many as 78% of children with autism spectrum disorder (ASD) have significant sleep disturbance compared to 20% of children without ASD. In children with ASD, shorter sleep duration and lower sleep efficiency, are associated with disruptive behavior, anxiety, and increased parental stress. Therefore, multiple sleep dimensions (B-SATED: behaviors, satisfaction, alertness, timing, efficiency, duration) are appropriate therapeutic targets to improve daytime behavioral functioning and other psychosocial outcomes. The primary objective is to evaluate the implementation of a modification of a behavioral sleep and circadian intervention to improve multiple sleep dimension in school-age children with ASD. To accomplish this objective, a 12-week, randomized pilot study will be conducted to assess the feasibility, acceptability, and preliminary efficacy of a modified behavioral sleep and circadian intervention with up to 50 school-age children with ASD, to determine whether the intervention improves multiple dimensions of sleep (B-SATED: behaviors, satisfaction, alertness, timing, efficiency, duration), daytime behavior, quality of life, parental stress, and parental self-efficacy.

This modified intervention is guided by the Pediatric Sleep Health Framework that encourages improvement in six pediatric sleep dimensions (B-SATED): sleep behaviors; parents' satisfaction with child sleep; daytime alertness/sleepiness; appropriate timing of sleep within the 24-hour day; sleep efficiency, i.e., ease of falling and staying asleep; and sleep duration. The Sadeh and Anders Sleep-Wake Regulation Model was used to propose linkages between outcomes. The investigators hypothesize that parents implementing the modified intervention will improve the primary outcome (clinician- and parent-ratings of child sleep) and secondary child (sleep dimensions, daytime behavior, quality of life) and parent outcomes (stress and self-efficacy).

DETAILED DESCRIPTION:
Study Overview: The overall goals are to adapt and evaluate the feasibility, acceptability, and preliminary efficacy of a modified behavioral sleep and circadian intervention for school-age children with autism spectrum disorder (ASD). Initial modifications were based on individual qualitative interviews with parents and feedback from a community advisory board to revise the existing intervention. A qualitative descriptive approach guided the modification of the intervention's content, format, delivery, and identification of barriers and facilitators. End-user feedback and debriefing were conducted with parents who participated in the qualitative interviews.

The final phase of the study involves conducting a randomized pilot study to assess the feasibility, acceptability, and preliminary efficacy of this intervention prototype. Our primary objective is to evaluate the implementation of a modified sleep and circadian intervention to improve multiple sleep dimensions in school-age children with ASD. To accomplish this objective, a 12-week, randomized pilot study will be conducted with up to 50 school-age children with ASD to assess the feasibility, acceptability, and preliminary efficacy of the intervention. The study aims to determine whether the intervention improves multiple dimensions of sleep (B-SATED: behaviors, satisfaction, alertness, timing, efficiency, duration), daytime behavior, quality of life, parental stress, and parental self-efficacy. The investigators hypothesize that parents implementing the modified intervention will improve the primary outcome (clinician- and parent-ratings of child sleep) and secondary child (sleep dimensions, daytime behavior, quality of life) and parent outcomes (stress and self-efficacy).

Study Design: A two-arm, RCT will be used to evaluate the preliminary efficacy, feasibility, and acceptability of the modified behavioral sleep intervention compared to a time-balanced attention control condition (enhanced usual care). Data collection will include T0 baseline measures (parent ratings and 7 nights of actigraphy sleep monitoring). After completing the baseline measures, participants will be allocated to either the experimental condition or the enhanced usual care control condition. T1 will include immediate post-intervention measures at 3 months (parent ratings and 7 nights of actigraphy sleep monitoring). T2 will include repeating measures at 6 months post-intervention (parent ratings only).

ELIGIBILITY:
Inclusion Criteria:

1. Children 6-12 years with a clinical diagnosis of ASD defined by the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition and corroborated by the Social Communication Questionnaire-lifetime score of ≥ 15.
2. Child must have ≥ 1 poor sleep health dimensions (B-SATED).
3. Child is not currently participating in any sleep-related interventions.
4. Child has not had any medication changes within the past month that interfere with sleep.
5. If present, the child must have a treated OSA (mild or less) diagnosis and willingness to continue treatment (≥80% adherence).
6. Parent must be an adult legal guardian proficient in English.

Exclusion Criteria:

1. Children with an untreated complex medical condition that interferes with sleep (e.g., epilepsy, nocturnal seizures).
2. Children with moderate to severe OSA.
3. Unable to complete protocol (e.g., serious behavioral concerns, bereavement, currently homeless).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The Improvement Scale of the Clinical Global Impressions Scale (CGI-I) | Baseline, Post-Intervention (Week 12), and Follow Up (Week 24)
  The improvement scale of Clinical Global Impression (CGI-I) Scale will be used to evaluate treatment-related improvement. The CGI-Improvement scale is rated by a clinician on a scale of 1 to 7, with 1 representing "very much improved" and 7 representing "very much worse." The CGI-Improvement scale (Scores 1 "very much improved" or 2 "much improved") will be used to identify a positive response to treatment.
Change in the Pediatric Autism Insomnia Rating Scale (PAIRS) | Baseline, Post-Intervention (Week 12), and Follow Up (Week 24)
  The PAIRS is a parent rating of insomnia and sleep-related impairments over the past two weeks in children with ASD age 3 to 12 years. The PAIRS is a single-factor measure comprising 21 items that assess difficulties with falling and/or staying asleep, as well as the impact of sleep problems on the child and the family. Items are scored: 0 (mild = not present, not a problem) to 3 (severe = frequent and a major problem). Higher scores indicate greater severity.

SECONDARY OUTCOMES:
Change in Child Sleep Dimensions Composite Score | Baseline, Post-Intervention (Week 12)
  Behaviors, Satisfaction, Alertness, Timing, Efficiency, Duration (B-SATED) sleep dimensions is a composite score that will be measured by the Modified Children's Sleep Habits Questionnaire (M-CSHQ), sleep diaries, and/or actigraphy [Poor sleep dimensions = Behaviors-M-CSHQ and sleep diary items related to bedtime routine consistency, sleep onset associations, co-sleeping, caffeine intake, and bedtime media use-endorsement of any of these items indicates poor sleep behaviors; Satisfaction-M-CSHQ total ≥ 33; Alertness/Sleepiness-M-CSHQ alertness score ≥ 10; Timing/Regularity-variability in bed/waketimes ≥ 1 hour; sleep Efficiency < 85%; sleep Duration < 9 hours per 24-hour period]. One overall score is derived from the six dimensions. Each dimension will be dichotomized as "1=good" or "0=poor" with scores ranging from 0-6, with a higher score indicating better sleep. Cutoffs are based on pediatric sleep recommendations.
Change in Child Daytime Behavior | Baseline, Post-Intervention (Week 12), and Follow Up (Week 24)
  The Aberrant Behavior Checklist (ABC) is a parent rating of child behavior with five subscales: Irritability (15 items), Lethargy/Social Withdrawal (16 items), Stereotypic Behavior (7 items), Hyperactivity/ Noncompliance (16 items), and Inappropriate Speech (4 items). The ABC consists of 58-items scored: 0 (never a problem) to 3 (severe problem). Higher scores indicate greater severity.
Change in Child Health-Related Quality of Life | Baseline, Post-Intervention (Week 12), and Follow Up (Week 24)
  The PedsQL 4.0 will be used to measure pediatric health-related quality of life (HRQoL). The 23-item PedsQL Generic Core Scale is used to measure pediatric HRQoL and covers four domains related to functioning: Physical (8 items), Emotional (5 items), Social (5 items), and School (5 items for children). Items are scored on a 5-point Likert-type scale (range, 0 = never a problem; 4 = almost always a problem). To compute summary scores, items are reversed scored and linearly transformed to a 0-100 scale. Higher scores indicate better pediatric HRQoL.
Change in Parental Stress | Baseline, Post-Intervention (Week 12), and Follow Up (Week 24)
  The Parenting Stress Index-Short Form (PSI-SF) is a 36-item tool specifically designed to measure parenting stress. Items are scored on a 5-point likert scale with 1 = strongly disagree and 5 = strongly agree. There are three subscales of the PSI-SF, each containing 12 items: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Total scores can range from 36 to 180. Higher scores indicate higher levels of parenting stress.
Change in Parental Sense of Competence | Baseline, Post-Intervention (Week 12), and Follow Up (Week 24)
  The Parenting Sense of Competence Scale (PSOC) consists of 17-items that are designed to measure parental satisfaction and self-efficacy. Items are scored on a 6-point scale with scores ranging from "strongly agree" = 6 to "strongly disagree" = 1. Higher scores reflect greater parental competence.
Change in Parental Sleep Quality | Baseline and Post-Intervention (Week 12)
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item questionnaire designed to assess sleep quality and disturbances. It evaluates seven components of sleep, which are combined to produce a global score ranging from 0 to 21. A total score of 5 or higher indicates clinically significant sleep difficulties, with higher scores reflecting poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Megan L Wenzell, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No